CLINICAL TRIAL: NCT01519908
Title: Markers and Response to Cardiac Resynchronization Therapy
Acronym: MARC
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Center for Translational Molecular Medicine (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other); Free University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CTMM-COHFAR-MARC
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy; biomarkers; response
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CRT-D (Medtronic) — Biventricular implantable cardioverter defibrillator, post marketing release
  Other Names: Medtronic CRT-D device

SUMMARY:
The purpose of this study is to investigate: the relation of a set of (bio)markers and response to Cardiac Resynchronization Therapy (CRT); the interrelationship as well as the potential predictive power of these (bio)markers on improvement and/or deterioration of cardiac function, cardiac geometry (reverse re-modeling during CRT) will be evaluated.

(Bio)markers include but are not limited to: collagen, genomic markers, molecular markers, electrocardiographic markers, echocardiographic markers, arrhythmogenic markers and markers for renal function: blood urea nitrogen (BUN), serum creatinine, glomerular filtration rate (GFR).

DETAILED DESCRIPTION:
Title

MARC (Markers And Response to CRT) - Prospective CRT study

Sponsor and study management

The MARC study is being sponsored by all participants of the COHFAR project as being defined in the COHFAR project agreement (Medtronic, UMCU, AMC, MUMC, VUMC, UMCG and ICIN). Study management will be done by Medtronic.

Purpose

To investigate the relation of a set of (bio)markers and response to Cardiac Resynchronization Therapy (CRT); the interrelationship as well as the potential predictive power of these (bio)markers on improvement and/or deterioration of cardiac function, cardiac geometry (reverse re-modeling during CRT) will be evaluated.

(Bio)markers include but are not limited to: collagen, genomic markers, molecular markers, electrocardiographic markers, echocardiographic markers, arrhythmogenic markers and markers for renal function: blood urea nitrogen (BUN), serum creatinine, glomerular filtration rate (GFR).

Design:

This is a multi-center, exploratory, prospective, interventional post-market release, non-randomized, study.

Medical device:

For reasons of uniform therapy delivery and homogeneity of (device diagnostic) study data, only Medtronic CRT-Defibrillator devices are used in this study with CareLink transmission functionality, OptiVol and Cardiac Compass report. Any commercially available leads can be used upon discretion of the investigator. All CRT-D devices and additional components (leads, programmer) incorporated in this study are CE-marked and market-released devices and used within the intended use of these devices.

Objectives:

Primary objective

• To investigate the relationship between a set of (bio)markers and response to cardiac resynchronization therapy (as measured by echocardiography) at 6 months.

Secondary objectives

* To investigate the relationship between a set of (bio)markers and response to cardiac resynchronization therapy (as measured by echocardiography) at 12 months
* To investigate the relationship between (bio)markers and atrial fibrillation during follow-up
* To investigate the relationship between (bio)markers and ventricular tachycardia/ fibrillation and/or appropriate shocks during follow-up
* To investigate the relationship between (bio)markers and reverse remodeling
* To relate baseline cardiac anatomy, function and mechanical dyssynchrony by cardiac MR and PET imaging in a subset of patients to CRT-response and to atrial and ventricular arrhythmias.

The biomarkers include:

* Genomics (while blood cells): candidate gene approach with micro-RNA's (analysis will be performed at the Genetics Core laboratory at study end. A inal list of micro-RNA's will be determined at study end).
* Blood markers (serum or plasma) are but not limited to: biomarkers of fibrosis, inflammation, cardiac damage, hemodynamic stress and extra-cardiac markers and will be analyzed at the Blood Biomarkers Core laboratory at study end.
* CMR Imaging at baseline for patients enrolled at the VUMC, AMC and UMCU investigational centers: function, anatomy, hemodynamics, global and local mechanical dyssynchrony assessment (tagged MR, CURE, torsion), Scar Imaging (DCE-MRI) will be measured.
* PET Imaging for patients enrolled at the VUMC, AMC and UMCU investigational centers: Perfusion (Adenosine), Innervation withHED tracer will be performed.
* Electrocardiography: Beat-to-beat Variability of Repolarization (BVR) / Short-Term Variability (STV) protocol
* Echocardiography: function and structure (including but not limited to LVEDD, LVESV, LVEDV, LVESVi, LVEF, MR, LVFT, IVMD, atrial volumina), in combination with electrocardiographic investigation: PA-TDI (P-wave duration). Echo 2D-Speckle Tracking: Radial Strain, Septal Rebound Stretch, standard deviation of Time to peak systolic Strain (final set of parameters will be determined at study end).
* Clinical parameters including among other coronary artery disease, Body Mass Index, gender, Myocardial Infarction at baseline.

All blood samples will be taken from peripheral venous blood and during implant also from the coronary sinus.

Additional prospective analysis:

* HF monitoring: intra-thoracic impedance (Optivol), patient activity, heart rate variability, Cardiac Compass arrhythmic episodes, continuously recorded through Carelink
* Electrical markers: arrhythmogenic markers (final list of markers to be determined at study end).
* Correlation of AT/AF episodes as detected by Carelink with baseline PA Tissue Doppler Imaging data.
* Correlation of echo strain measurements and MRI strain measurements
* Occurrence of clinical events during long-term follow-up; clinical events include:

  * Cardiovascular hospitalizations
  * Heart failure hospitalizations
  * All-cause mortality
  * Heart transplantation
  * Acute implantation of a left ventricular assist device
  * Atrial and ventricular arrhythmias including atrial fibrillation, atrial flutter, atrial tachycardia, ventricular tachycardia, ventricular fibrillation, as documented by continuous device diagnostic monitoring through CareLink

Subject selection:

The study will enroll 240 symptomatic heart failure patients (NYHA functional class II-III) with a reduced left ventricular ejection fraction and a prolonged QRS duration as measured prior to implantation of a cardiac resynchronization device (CRT-D). All patients will be followed for 1 year after implant. Each patient will visit the clinical site at baseline, 1-month, 6-month and 12 month follow-up. The total study duration will be 3 years. The 5 participating clinical institutions are all located in the Netherlands and member of the COHFAR project which is a partnership of the Center for Translational Molecular Medicine (CTMM) and Universitair Medisch Centrum Utrecht (UMCU), Universitair Medisch Centrum Groningen (UMCG), Academisch Medisch Centrum (AMC), VU Medisch Centrum (VUMC), Maastricht Universitair Medisch Centrum (MUMC), Medtronic and MSD with support from the Dutch Heart Foundation.

Treatment:

Each study subject will receive cardiac resynchronization therapy (CRT-D) according to the ESC/AHA guidelines and per local hospital routine. Additionally, optimal medical therapy for heart failure is up to the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for CRT-D device according to current applicable ESC/AHA guidelines
* Subject has NYHA class II or III
* Subject has stable sinus rhythm (no atrial arrhythmias lasting > 30 seconds during the last 2 weeks prior to inclusion) No documented AF-episodes allowed during the last 2 weeks prior to inclusion.
* Intrinsic QRS-width ≥ 130 ms with LBBB or ≥ 150 ms without LBBB as measured within 30 days prior to device implant for subjects with NYHA class II
* Intrinsic QRS-width ≥ 120 ms with LBBB or ≥ 150 ms without LBBB as measured within 30 days prior to device implant for subjects with NYHA class III
* Subject receives optimal heart failure oral medical therapy (ACE inhibitor and/or ARB and Beta Blockers), and is on a stable medication scheme for at least 1 month prior to enrollment
* Subject is willing to sign informed consent form
* Subject is 18 years or older

Exclusion Criteria:

* Subject is upgraded from a bradycardia pacemaker to CRT-D
* Subject receives CRT-D replacement or is upgraded from CRT-P to CRT-D
* Subject has permanent atrial fibrillation/ flutter or tachycardia.
* Subject experienced recent myocardial infarction (MI), within 40 days prior to enrollment
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year
* Subject is implanted with a left ventricular assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year
* Subject is on chronic renal dialysis
* Subject has severe renal disease (defined as Glomerular Filtration Rate (GFR) < 30 mL/min/1.73m2)
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure (≥ 2 stable infusions per week)
* Subject has RBBB
* Subject has permanent 2nd or 3rd degree AV-block
* Subject has severe aortic stenosis (with a valve area of < 1.0 cm2 or significant valve disease expected to be operated within study period)
* Subject has complex and uncorrected congenital heart disease
* Subject has a mechanical right heart valve
* Subject has a life expectancy of less than one year in the opinion of the investigator
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Subject is enrolled in one or more concurrent studies that would confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group to be recruited will consist of symptomatic heart failure patients (NYHA II-III), male and female, with a reduced left ventricular ejection fraction and ventricular dyssynchrony as measured prior to implantation of a cardiac resynchronization therapy device (CRT-D). Each study subject receives a CRT-Daccording to the current ESC/AHA guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarkers with reverse remodeling in cardiac resynchronization therapy | 6 months
  To investigate the relationship between a set of (bio)markers and response to cardiac resynchronization therapy (as measured by echocardiography) at 6 months.
  For each biomarker, the relation with LVESVi change between baseline and 6 months post implant will be analyzed.

SECONDARY OUTCOMES:
Correlation of biomarker with reverse remodeling in cardiac resynchronization therapy | 12 months
  Secondary objective 1
  • To investigate the relationship between a set of (bio)markers and response to cardiac resynchronization therapy (as measured by echocardiography) at 12 months For each biomarker, the relation with LVESVi change between baseline and 12 months will be analyzed. This is identical to the primary objective, except that a 12 months horizon is used instead of 6 months.
Correlation of biomarkers and atrial fibrillation in cardiac resynchronization therapy | 12 months
  Secondary objective 2
  • To investigate the relationship between (bio)markers and atrial fibrillation during follow-up The purpose of this objective is to investigate if biomarkers can identify patients that have increased risk to get AF episodes, and to investigate if biomarkers can predict the amount of AF.
Correlation of biomarkers and ventricular arrhythmias in cardiac resynchronization therapy | 12 months
  Secondary objective 3
  • To investigate the relationship between (bio)markers and ventricular tachycardia/ fibrillation and/or appropriate shocks during follow-up The purpose of this objective is to investigate if biomarkers can identify patients that have increased risk to get VF episodes.
Correlation of biomarkers with echocardiographic changes in cardiac resynchronization therapy | 12 months
  Secondary objective 4
  • To investigate the relationship between (bio)markers and reverse remodeling The primary objective will look at change of LVESVi. The purpose of this secondary objective is to confirm results of the primary objective by looking at other cardiac volume and dimension measurements, including LVESV, LVEDV and LVEDD.
Correlation of anatomy and function with response to cardiac resynchronization therapy | 12 months
  Secondary objective 5
  • To relate baseline cardiac anatomy, function and mechanical dyssynchrony by cardiac MRI and PET imaging in a subset of patients to CRT-response and to atrial and ventricular arrhythmia's.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vos, MD, PhD, Study Director — UMC Utrecht
Locations (6):
- Netherlands (6):
  - Academic Medical Center, Amsterdam
  - Free University, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Salden OAE, Zweerink A, Wouters P, Allaart CP, Geelhoed B, de Lange FJ, Maass AH, Rienstra M, Vernooy K, Vos MA, Meine M, Prinzen FW, Cramer MJ. The value of septal rebound stretch analysis for the prediction of volumetric response to cardiac resynchronization therapy. Eur Heart J Cardiovasc Imaging. 2021 Jan 1;22(1):37-45. doi: 10.1093/ehjci/jeaa190. PMID 32699908
- [Derived] Maass AH, Vernooy K, Wijers SC, van 't Sant J, Cramer MJ, Meine M, Allaart CP, De Lange FJ, Prinzen FW, Gerritse B, Erdtsieck E, Scheerder COS, Hill MRS, Scholten M, Kloosterman M, Ter Horst IAH, Voors AA, Vos MA, Rienstra M, Van Gelder IC. Refining success of cardiac resynchronization therapy using a simple score predicting the amount of reverse ventricular remodelling: results from the Markers and Response to CRT (MARC) study. Europace. 2018 Feb 1;20(2):e1-e10. doi: 10.1093/europace/euw445. PMID 28339818
- See also: Related Info — http://www.ctmm.nl